CLINICAL TRIAL: NCT04430062
Title: Short-term Outcome of Covid-19 Surgical Patients: Case-series of a High-risk Area Community Hospital
Status: Completed | Type: Observational
Sponsor: Azienda Socio Sanitaria Territoriale di Lodi (Other)
Responsible Party: Principal Investigator, Michele Ballabio, Michele Ballabio, MD, Principal Investigator, Azienda Socio Sanitaria Territoriale di Lodi
Other Study IDs: Covid19nr1
Record Dates: First submitted 2020-06-11; First posted 2020-06-12 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: General Surgery; Disease Outbreaks
Keywords: Surgery; Covid-19; SARS-CoV-2; Surgical outcome
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid-19 patients operated (February 21st -April 10th)
  Interventions: Procedure: Surgical procedures performed under general anesthesia

INTERVENTIONS:
Procedure: Surgical procedures performed under general anesthesia — Surgical procedures performed under general anesthesia in patients with perioperative SARS-CoV-2 infection

SUMMARY:
The investigators retrospectively evaluated all the patients operated in a high-risk community hospital from the first Italian case of Covid-19 (February 21st) to the April 10th (in order to have at least a 30-days follow-up). The investigators selected those patients who had a preoperative or post-operative positive Real Time - Polymerase Chain Reaction (RT-PCR) for SARS-CoV-2 and the clinical outcome of the participants was evaluated in term of need of Intensive Care Unit (ICU) post-operative recovery, medical and surgical complications, length of hospital stay and death.

ELIGIBILITY:
Inclusion Criteria:

* preoperative or post-operative positive Real Time - Polymerase Chain Reaction (RT-PCR) for SARS-CoV-2
* surgical procedure in elective or acute care surgery performed under general anesthesia

Exclusion Criteria:

* patients operated without general anesthesia
* patients preoperatively intubated for Covid-19

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: General population referring to a community hospital during the SARS-CoV-2 outbreak in the Northern Italy
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale di Lodi - ASST Lodi, Lodi, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No